CLINICAL TRIAL: NCT03188289
Title: Randomized Clinical Trial of Microbial Growth in the Suture Thread, After the Post-surgical Application of Different Antiseptic Gels in Mandibular Third Molars Extraction
Brief Title: Microbial Growth in the Suture Thread, After Application of Different Antiseptic Gels in Mandibular Third Molars Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Samuel Rodríguez Zorrilla, DDS, MSc., University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2017-05-28; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Wisdom Teeth; Oral Surgery; Third Molar Surgery; Bioadhesive Gel; Suture Bacteria; Antiseptic Gel; Chistosan; Clorhexidine Gel Bacteria; Clorhexidine-chitosan; Bacterial Growth
Keywords: chitosan; clorhexidine; suture; bacteria; wisdom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo gel (Placebo Comparator): The placebo gel is used by all patients on one side of the mouth and serves as a control group.
  Interventions: Drug: Placebo gel; Drug: Clorhexidine gel; Drug: Clorhexidine-Chitosan gel; Drug: Hyaluronic Acid gel
- Clorhexidine gel (Active Comparator): Chlorhexidine gel is one of three gels used to compare the placebo gel and will be used on the contralateral side to the side assigned as placebo in a third of the participants.
  Interventions: Drug: Placebo gel; Drug: Clorhexidine gel; Drug: Clorhexidine-Chitosan gel; Drug: Hyaluronic Acid gel
- Clorhexidine-Chitosan gel (Active Comparator): Clorhexidine-chitosan gel is one of three gels used to compare the placebo gel and will be used on the contralateral side to the side assigned as placebo in a third of the participants.
  Interventions: Drug: Placebo gel; Drug: Clorhexidine gel; Drug: Clorhexidine-Chitosan gel; Drug: Hyaluronic Acid gel
- Hyaluronic acid gel (Active Comparator): Hialuronic acid gel is one of three gels used to compare the placebo gel and will be used on the contralateral side to the side assigned as placebo in a third of the participants.
  Interventions: Drug: Placebo gel; Drug: Clorhexidine gel; Drug: Clorhexidine-Chitosan gel; Drug: Hyaluronic Acid gel

INTERVENTIONS:
Drug: Placebo gel — Placebo is the control group treated with a placebo gel.
  Other Names: Hyspagel 200
Drug: Clorhexidine gel — Clorhexidine will be compare with placebo, clorhexidine-chitosán and hyaluronic acid bioadhesive gels
  Other Names: Bexident encías
Drug: Clorhexidine-Chitosan gel — Clorhexidine-chitosan will be compare with placebo, clorhexidine and hyaluronic acid bioadhesive gels.
  Other Names: Bexident Post
Drug: Hyaluronic Acid gel — Hyaluronic acid will be compare with placebo, clorhexidine, clorhexidine-chitosan bioadhesive gels
  Other Names: Oddent

SUMMARY:
This is a randomized clinical trial in which investigators will compare the antimicrobial effect and inducer of cicatrization as well as the degree of postoperative pain in patients who are extracted the lower third molars.

After the surgery, different bioadhesive gels will be applied in the area of the surgical wound and we will evaluate the aforementioned parameters.

DETAILED DESCRIPTION:
Introduction: Surgical removal of the third molars is one of the most frequent procedures in oral surgery. Healing of the wound is initially sought by approximating the edges using a suturing technique. Adherence and microbiological accumulation of the suture during the period that it remains in the mouth, which can serve as a focus for odontogenic infections. The use of oral antiseptics before and after the surgery is an efficient method for microbial reduction. The purposes of this project were to evaluate the microbial growth in the suture thread on different culture means after the post-surgical application of the gels under study, while assessing the intensity of post-surgical pain and the degree of healing of the surgical wound.

Material and methods: It is a randomized and blind clinical trial. 21 patients participated (42 wisdom teeth), who consulted the unit for a surgical tooth extraction for at least the two lower wisdom teeth. The evaluated bioadhesive gels were: Chlorhexidine gel at 0.2 % (Bexident Gel Gingival®), Chlorhexidine gel at 0.2% + Chitosan (Bexident Post®) and hyaluronic acid gel (ODDENT®). A neutral water-based gel without any active ingredients was also used HISPAGEL 200® (Acofarma, Madrid, Spain) as the control agent. An assessment of the post-surgical healing, the microbiological analysis of the suture thread and the post-surgical pain was developed.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 39 years.
* Good general health.
* Availability during the study.
* No current odontological treatments or foreseen during the study period.
* Acceptance and compliance with the prescribed oral hygiene instructions.
* Agreement to not used mouthwashes or toothpastes with antiseptic agents during the study period.

Exclusion Criteria:

* Use of antimicrobial mouthwashes or toothpastes during the period during which the suture remains in the mouth.
* Diabetes.
* Smoking.
* Degenerative diseases.
* Deficient oral health (cavities, periodontal disease, pathologies of the oral mucosa...).
* Wearing prosthetic or orthodontic devices.
* Amoxicillin allergy.
* Pregnant or lactating women.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2014-07-15 (Actual); Study Completion 2014-09-10 (Actual)

PRIMARY OUTCOMES:
Microbiological growth on suture tread. | Seven days.
  Microbiological growth in CFUs on the suture thread after the application of the distinct bioadhesive gels.
Postoperative pain in the operated area. | Seven days.
  The researchers will analyze the degree of postoperative pain patients suffered during the first postoperative week by applying one of the gels to be studied in the area of the surgical wound. To make this measurement the visual analogue pain scale will be used.
Degree of healing. | Seven days.
  The degree of healing at 7 days after surgery was measured using a visual healing scale consisting of four different levels of healing status:
  1. - Erithymatous surgical zone and with signs of inflammation and infection.
  2. - Erythematous surgical site without signs of infection.
  3. -Surgical zone of normal color and beginning of epithelization.
  4. -Surgical zone of normal color and advanced epithelization.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Rodríguez Zorrilla, DDS,MSc, Principal Investigator — University of Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No